CLINICAL TRIAL: NCT02141061
Title: A Double-Blind Crossover Study in Healthy Volunteers to Compare Two Formulations of Proellex for Oral Administration
Brief Title: Comparison of Two Formulations of Proellex for Oral Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: ZPU-101
Record Dates: First submitted 2014-05-13; First posted 2014-05-19 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telapristone Acetate, Proellex Formulation A (Treatment A) (Experimental): Subjects who meet the eligibility criteria will be randomized to receive either 12 mg Treatment A or 12 mg Treatment B as their first assigned treatment. After a 7-day washout period subjects will receive the alternative treatment.
  Interventions: Drug: Telapristone Acetate, Proellex 12 mg Formulation A; Drug: Telapristone Acetate, Proellex 12 mg Formulation B
- Telapristone Acetate, Proellex Formulation B (Treatment B) (Experimental): Subjects who meet the eligibility criteria will be randomized to receive either 12 mg Treatment A or 12 mg Treatment B as their first assigned treatment. After a 7-day washout period subjects will receive the alternative treatment.
  Interventions: Drug: Telapristone Acetate, Proellex 12 mg Formulation A; Drug: Telapristone Acetate, Proellex 12 mg Formulation B

INTERVENTIONS:
Drug: Telapristone Acetate, Proellex 12 mg Formulation A
  Other Names: Proellex
Drug: Telapristone Acetate, Proellex 12 mg Formulation B
  Other Names: Proellex

SUMMARY:
This study is a double-blind crossover study in female healthy volunteers to compare the pharmacokinetics and safety of a single dose each of two different formulations of Proellex for oral administration. Each formulation will be designated as either Treatment A or Treatment B. A total of 12 subjects who meet the eligibility criteria will be randomized to receive either Treatment A or Treatment B as their first assigned treatment. After a 7-day washout period subjects will receive the alternative treatment. On the day of each treatment subjects will remain in the clinic overnight and undergo 72-hour pharmacokinetic assessment at the following time points: 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48 and 72 hours after administration of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an IRB-approved form prior to the initiation of any study procedures;
2. Healthy, premenopausal female age 18-47;
3. History of menstrual events that occur in regular cycles
4. Agreement not to attempt to become pregnant
5. Agrees to use double-barrier contraception during the study and for 30 days after discontinuation of study medication. Acceptable double-barrier methods are: male condom with spermicide; male condom with diaphragm; diaphragm containing spermicide plus additional intra-vaginal spermicide;
6. Has a negative pregnancy test at the Screening visit. An exception for the pregnancy test requirement will be granted for subjects reporting surgical sterilization in medical history
7. Normal laboratory values or clinically insignificant findings at screening as determined by the Investigator;
8. Subject is willing to remain in the clinic overnight for PK assessment on Days 0 and 8
9. Ability to complete the study procedures in compliance with the protocol.

Exclusion Criteria:

1. Subject is a post-menopausal woman, defined as either; six (6) months or more (immediately prior to screening visit) without a menstrual period, or prior hysterectomy and/or oophorectomy
2. Subject is pregnant or lactating or is attempting or expecting to become pregnant during the study
3. Women with abnormally high liver enzymes or liver disease. (ALT or AST exceeding 2.0 x ULN AND total bilirubin exceeding 1.5 x ULN at screening and confirmed on repeat).
4. Received an investigational drug in the 30 days prior to the screening for this study
5. Women with a history of PCOS
6. Concurrent use of any testosterone, progestin, androgen, estrogen, anabolic steroids, DHEA or hormonal products for at least 2 weeks prior to screening and during the study.
7. Use of oral contraceptives in the preceding 2 weeks. Use of Depo-Provera® in the preceding 10 months.
8. Has an IUD in place
9. Women currently using narcotics
10. Women currently taking spironolactone
11. Infectious disease screen is positive for HIV or Hepatitis A, B or C.
12. Clinically significant abnormal findings on screening examination or any condition which in the opinion of the investigator would interfere with the participant's ability to comply with the study instructions or endanger the participant if she took part in the study

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Comparison | Up to 2 weeks
  To determine and compare the pharmacokinetics (PK) of a single dose of each of two formulations of 12 mg Proellex administered orally to female healthy volunteers. On the day of each treatment subjects will remain in the clinic overnight and undergo 72-hour pharmacokinetic assessment at the following time points: 0, 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48 and 72 hours after administration of study drug.
  Pharmacokinetic Endpoints
  * AUC 0-t
  * AUC 0-24
  * AUC 0-∞
  * Cmax
  * Tmax
  * λz
  * t½
Dose formulation safety | Up to 2 weeks
  To determine and compare the safety of a single dose of each of two formulations of 12 mg Proellex administered orally to female healthy volunteers. After the completion of the study; incidence of adverse events, mean change from baseline of laboratory values (hematology, blood chemistry, urinalysis), mean change from baseline of vital signs will be assessed. Vital signs and adverse events will be recorded at each visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Houston, Texas, United States